CLINICAL TRIAL: NCT05716659
Title: Assessment of Brain-heart-muscle Axis Using EEG/MECG/EMG Combo Machine for Evaluating the Severity of Aortic Stenosis, Heart Failure and Ischemic Stroke Through an Artificial Intelligenceassisted System.
Brief Title: EEG/MECG/EMG Evaluating the Severity of Aortic Stenosis, Heart Failure and Ischemic Stroke Through an Artificial Intelligenceassisted System.
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202207146DIPB
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2022-12

CONDITIONS: CVD
Keywords: heart failure; aortic stenosis; ischemic stroke
MeSH Terms: conditions — Heart Failure; Aortic Valve Stenosis; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Healthy subjects group: 150 healthy subjects
- Metabolic syndrome group: 100 patients with clinical diagnosis of metabolic syndrome.
- Heart failure group: 100 patients with clinical diagnosis of heart failure.
- Heart failure with metabolic syndrome group: 100 patients with clinical diagnosis of heart failure with metabolic syndrome.
- Severe aortic valve stenosis group: 100 patients with clinical diagnosis of severe aortic valve stenosis.
- Ischemic stroke group: 200 patients with clinical diagnosis of ischemic stroke.

SUMMARY:
The specific objectives and methods of this project are: (1) To test the feasibility and accuracy of integrating EEG, MECG and EMG for detecting the severity of diseases such as aortic stenosis, heart failure and ischemic stroke. (2) Improve the accuracy of this multi-channel brain-heart-muscle device by using an artificial intelligence auxiliary system. (3) Provide tailor-made interdisciplinary treatment strategies for patients with different disease states.

ELIGIBILITY:
Inclusion criteria

1. Age≥20 year-old
2. Healthy subjects or patients with A. Metabolic syndrome (MetS) ；B. HF with reduced ejection fractions (HFrEF, defined by left ventricular ejection fraction≤40%) and current or previous symptoms of HF；C. Severe aortic stenosis (defined aortic valve area < 1.0 cm2 or mean pressure gradient ≥ 40 mmHg), preparing to receive transcatheter aortic valve replacement ；D. Acute ischemic stroke and admitted to stroke intensive care unit (ICU), within 24 hours after onset

The criteria of MetS includes:

1. Abdominal obesity: waist circumference (for Asians) ≥ 90 cm in men and ≥ 80 cm in women;
2. Hyperglycemia: serum fasting glucose level ≥ 100 mg/dl, or receiving drug treatment for elevated blood sugar;
3. Reduced high-density lipoprotein cholesterol (HDL-C): serum HDL-C < 40 mg/dl in men and < 50 mg/dl in women or on cholesterol drug treatment;
4. Elevated triglycerides: serum triglyceride ≥ 150 mg/dl or on drug treatment of hypertriglyceridemia;
5. Hypertension: systolic blood pressure ≥ 130 mmHg, diastolic blood pressure ≥ 85 mmHg, or on antihypertensive drug treatment.

Exclusion criteria:

1. Under treatment for malignancy
2. Currently receiving immunosuppressants
3. Modified Rankin Scale (mRS) ≥2 prior to the stroke
4. Symptomatic HF in patients with acute ischemic stroke
5. Unable to perform neurocognitive function test
6. Unable to evaluate the physical activity using questionnaire or 6-minute walk test
7. Unable to cooperate with examinations using 3E combo machine.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this project, seven hundred and fifty male or female patients with healthy subjects or meet the inclusion conditions of the following four diseases over 20 years of age will be enrolled.
  A. Patients with metabolic syndrome
  B. Patients with heart failure
  C. Patients with severe aortic valve stenosis who have been evaluated as suitable for transcatheter aortic valve replacement
  D. Acute ischemic stroke patients admitted to stroke intensive care unit
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2032-07-31 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
Composite cardiovascular outcome | up to 10 years
  Composite endpoint: Major adverse cardiac events (MACE): myocardial infarction, stroke, hospitalization for heart failure, or cardiovascular death)

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Li Kao, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No